CLINICAL TRIAL: NCT02389725
Title: The Effect of Two Different Tourniquet Techniques on Peripheral IV Access Success Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Tobias Kummer, Assistant Professor of Emergency Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 14-007501
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Results first posted 2019-05-20 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-04

CONDITIONS: Tourniquet
Keywords: peripheral intravenous access; tourniquet techniques

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- disposable elastic tourniquet (Active Comparator)
  Interventions: Device: disposable elastic tourniquet
- manual blood pressure cuff (Active Comparator): manual blood pressure cuff inflated to 150 milliliters mercury (mmHg)
  Interventions: Device: blood pressure cuff

INTERVENTIONS:
Device: disposable elastic tourniquet — Comparison of first time peripheral IV access success rate between the standard elastic tourniquet and a blood pressure cuff.
  Arms: disposable elastic tourniquet
Device: blood pressure cuff — Comparison of first time peripheral IV access success rate between the standard elastic tourniquet and a blood pressure cuff.
  Arms: manual blood pressure cuff

SUMMARY:
The purpose of this study is to compare the success rates of two different tourniquets that are used when placing an IV.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Department patients
* 18 years old or older
* who receive peripheral IV access

Exclusion Criteria:

* Patients under the age of 18
* prison inmates
* pregnant patients
* patients who are unable to give informed consent
* critically ill patients who need emergent IV access as defined by the Emergency Medicine consultant of record for the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Kummer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Result] Tran T, Lund SB, Nichols MD, Kummer T. Effect of two tourniquet techniques on peripheral intravenous cannulation success: A randomized controlled trial. Am J Emerg Med. 2019 Dec;37(12):2209-2214. doi: 10.1016/j.ajem.2019.03.034. Epub 2019 Mar 23. PMID 30948254
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Disposable Elastic Tourniquet | Manual Blood Pressure Cuff
Started | 59 | 60
Completed | 59 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Disposable Elastic Tourniquet | Manual Blood Pressure Cuff | Total
Number analyzed (Participants) | 59 | 60 | 119
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67 [54 to 78] | 62 [41 to 75] | 65 [46 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 35 | 68
  Male | 26 | 25 | 51
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 59 | 60 | 119

OUTCOME MEASURES:

1. Primary Outcome: Peripheral IV Access Success Rate
Description: Peripheral IV access success rate is defined as the number of subjects who had successful peripheral intravenous cannulation on the first attempt. An attempt was defined as a needle penetrating the surface of the subject's skin. Successful access was defined as good flow through an IV catheter with a saline flush and without subcutaneous fluid collection.
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Disposable Elastic Tourniquet | Manual Blood Pressure Cuff
Number analyzed (Participants) | 59 | 60
Participants | 42 | 43
Statistical Analysis 1: Comparison: Disposable Elastic Tourniquet vs Manual Blood Pressure Cuff; Test type: Superiority; p = 0.95, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Total Number of Peripheral IV Access Attempts
Description: The total number of peripheral IV access attempts for each subject., up to a maximum of four attempts. An attempt is defined as a needle penetrating the subject's skin surface.
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Groups:
- Manual Blood Pressure Cuff: manual blood pressure cuff inflated to 150mm Hg
Arm/Group | Disposable Elastic Tourniquet | Manual Blood Pressure Cuff
Number analyzed (Participants) | 59 | 60
Participants
  One attempt | 42 | 43
  Two attempts | 13 | 9
  Three attempts | 3 | 6
  Four attempts | 1 | 2
Statistical Analysis 1: Comparison: Disposable Elastic Tourniquet vs Manual Blood Pressure Cuff; Test type: Superiority; p = 0.87, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Total Number of Distinct Providers That Attempted IV Access
Description: Total number of individual medical providers that attempt to access IV for each subject. An attempt is defined as a needle penetrating the surface of the subject's skin. Access was defined as good flow through an IV catheter with a saline flush and without subcutaneous fluid collection.
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Disposable Elastic Tourniquet | Manual Blood Pressure Cuff
Number analyzed (Participants) | 59 | 60
Participants
  One provider | 51 | 50
  Two providers | 7 | 10
  Three providers | 1 | 0
Statistical Analysis 1: Comparison: Disposable Elastic Tourniquet vs Manual Blood Pressure Cuff; Test type: Superiority; p = 0.67, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Rate of Rescue Techniques Used
Description: The number of subjects requiring one or more rescue techniques to access peripheral IV. These techniques include ultrasound guided peripheral IV access, central venous access, venous cut-down, interosseous access, and/or change in treatment plan due to unsuccessful access.
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Groups:
- Manual Blood Pressure Cuff: manual blood pressure cuff inflated to 150 milliliters mercury (mmHg)
  .
Arm/Group | Disposable Elastic Tourniquet | Manual Blood Pressure Cuff
Number analyzed (Participants) | 59 | 60
Participants | 6 | 3
Statistical Analysis 1: Comparison: Disposable Elastic Tourniquet vs Manual Blood Pressure Cuff; Test type: Superiority; p = 0.32, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the duration of the IV placement during the emergency department visit, approximately 45 minutes.
Arm/Group | Disposable Elastic Tourniquet | Manual Blood Pressure Cuff
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/60
Other Adverse Events (participants affected / at risk) | 0/59 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes